CLINICAL TRIAL: NCT05250336
Title: Prognostic and Predictive Value of Tumor-Infiltrating Lymphocytes and Programmed Cell Death - Ligand 1 in Breast Cancer
Brief Title: Tumor-Infiltrating Lymphocytes and Programmed Cell Death - Ligand 1 in Breast Cancer
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Sanjay Gandhi Postgraduate Institute of Medical Sciences (Other Government)
Responsible Party: Principal Investigator, Gaurav Agarwal, Professor of Endocrine and Breast Surgery, Sanjay Gandhi Postgraduate Institute of Medical Sciences
Other Study IDs: 2018-177-IMP-EXP-4
Record Dates: First submitted 2022-02-11; First posted 2022-02-22 (Actual); Last update posted 2022-02-22 (Actual); Status verified 2022-02

CONDITIONS: Breast Cancer; Tumor Infiltrating Lymphocytes; Programmed Cell Death Ligand 1
MeSH Terms: conditions — Breast Neoplasms | interventions — Observation

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Other
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Patients with Primary Breast Cancer: The pretherapeutic cores or specimen from patients who meet the following criteria were subjected for analysis
  INCLUSION CRITERIA Primary Breast cancer Completed scheduled treatment at SGPGI Adequate quality histopathology material available in Department of Pathology archives With minimum 6 months follow up
  EXCLUSION CRITERIA Insufficient data Incomplete treatment Insufficient follow up information Insufficient histological material for review
  Interventions: Other: Observational Study

INTERVENTIONS:
Other: Observational Study — Assessment of Prognostic and Predictive value of Tumor-Infiltrating Lymphocytes and Programmed cell Death - Ligand 1 in Breast cancer

SUMMARY:
The morphological evaluation of Tumor-infiltrating Lymphocytes (TILs) in breast cancer is gaining momentum as evidence strengthens for the clinical relevance of this immunological biomarker. In breast cancer (BC) lesions, TILs are seen in intratumoral and stromal areas. TILs are predictive of response to treatment and this association appears to be strongest in Triple-negative (TNBC) and Her 2 (Human epidermal growth factor receptor) positive breast cancer subtypes. Contrastingly, the association in Estrogen Receptor (ER) positive, HER 2 negative tumors have not been established.

Programmed cell death 1 (PD-1), are receptors expressed on the surface of T, B, and Natural killer cells and in some tumor cells. These attenuate the cellular immune response by inducing T-cell apoptosis. Programmed Cell Death Ligand 1 (PD-L1) overexpression is reported to be associated with large tumor size, lymph node metastasis, and ER-negativity. Importantly, PD-L1 is expressed more frequently in TNBC patients. High PD-L1 expression may be a prognostic indicator for reduced overall survival6. This information may be helpful to screen candidates for anti-PD-1/PD-L1 therapy, especially patients with TNBC The aim of this study is to characterize the cohort of patients with breast cancer based on a semiquantitative assessment of TILs and to correlate the concentration of TILs and PD-L1 in various intrinsic subtypes (based on Immunohistochemistry) with the overall outcome. Also to correlate the TILs and PD-L1 expression with tumor response to Neoadjuvant Chemotherapy (NACT) and to stratify the predictive value of this biomarker in TNBC.

DETAILED DESCRIPTION:
This is a retrospective and prospective study in patients with Primary Breast cancer at Sanjay Gandhi Postgraduate Institute of Medical Sciences (SGPGI). This is a time-bound study, where we include all patients treated between January 2016 and December 2021 who meet the inclusion criteria. We screened out approximately 2000 patients treated over this period, of which about 1000 had met inclusion criteria.

The electronic and physical records of all breast cancer patients maintained in Hospital Information System and Department of Breast and Endocrine Surgery at SGPGI have been screened to identify all appropriate cases and their clinical data were reviewed.

The cohort of patients who met the inclusion criteria was identified from the screened data.

The paraffin blocks of pre-therapeutic core biopsies/ surgical specimens of the study subjects were retrieved and the same from prospective study subjects were included.

Existing data on Immunohistochemistry (IHC) for ER (Estrogen Receptor), PR (Progesterone Receptor), Her 2 neu (Human epidermal growth factor receptor) was tabulated to identify TNBC cohort.

Hematoxylin & Eosin stained histological slides were reviewed by one set of pathologists for semi quantification of TILs.

TILs have been analyzed both as continuous parameters and in three predefined groups of Low: 0-10%; Intermediate:11 - 59 % and high: ≥ 60 % stromal TILs. In patients with TNBC, the paraffin blocks were retrieved and PD-L1 expression was assessed by IHC.

At this point in time, the recruitment of subjects and semi-quantification of TILs and PDL-1 were over and the analysis/correlation part is yet to be done.

In all study subjects, the concentration of TILs will be correlated with the clinicopathological outcome (treatment response, overall survival, disease-free survival ) and this association will be compared between intrinsic subtypes based on IHC.

In patients treated with Neoadjuvant Chemotherapy (NACT), correlation of TILs with response to NACT (pathologic complete response, partial/static/progression) will be done.

Correlation of PDL-1 expression with outcomes (overall survival, disease-free survival) and with response to Neoadjuvant Chemotherapy (pathologic complete response, partial/static/progression) in patients with Triple Negative Breast Cancer will be done.

The study information obtained will be statistically analyzed to identify the significance of the aforementioned correlations.

ELIGIBILITY:
Inclusion Criteria:

* Primary Breast cancer
* Completed scheduled treatment at SGPGI
* Adequate quality histopathology material available in Department of Pathology archives
* With minimum 6 months follow up

Exclusion Criteria:

* Insufficient data
* Incomplete treatment
* Insufficient follow up information
* Insufficient histological material for review

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: This is a time-bound study, where we include all patients treated between January 2016 and December 2021 who meet the inclusion criteria.
  We had screened out approximately 2000 patients treated over this period, of which about 1000 have met the inclusion criteria.
Sampling Method: Non-Probability Sample
Enrollment: 1000 (Estimated)
Dates: Start 2019-01-19 (Actual); Primary Completion 2022-06-30 (Estimated); Study Completion 2022-09-30 (Estimated)

PRIMARY OUTCOMES:
Correlation of TILs and PDL-1 in various molecular sub-types | Range of 6 months - 6 years follow up
  To Correlate the concentration of TILs and PD-L1 in various intrinsic subtypes (based on Immunohistochemistry) with the overall outcome
PDL-1 expression in patients with Triple Negative Breast Cancer (TNBC) | a follow up period of 6 months to 6 years
  To Correlate PDL-1 expression with outcomes in patients with TNBC
TILs and Tumor response to treatment | a follow-up time frame Range from 6 months to 6 years
  To Correlate the TILs with tumor response to Neoadjuvant Chemotherapy and to stratify the predictive value of this biomarker
PD-L1 expression and Tumor response to treatment | Time frame range of 6 months to 6 years follow up
  To Correlate PD-L1 expression with response to Neoadjuvant Chemotherapy in patients with TNBC

CONTACTS AND LOCATIONS:
Overall Officials: Gaurav Agarwal, Principal Investigator — Sanjay Gandhi Postgraduate Institute of Medical Sciences, Lucknow, India
Locations (1):
- Sanjay Gandhi Postgraduate Institute of Medical Sciences, Lucknow, Uttar Pradesh, India

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Wein L, Savas P, Luen SJ, Virassamy B, Salgado R, Loi S. Clinical Validity and Utility of Tumor-Infiltrating Lymphocytes in Routine Clinical Practice for Breast Cancer Patients: Current and Future Directions. Front Oncol. 2017 Aug 3;7:156. doi: 10.3389/fonc.2017.00156. eCollection 2017. PMID 28824872
- [Background] Loi S, Michiels S, Salgado R, Sirtaine N, Jose V, Fumagalli D, Kellokumpu-Lehtinen PL, Bono P, Kataja V, Desmedt C, Piccart MJ, Loibl S, Denkert C, Smyth MJ, Joensuu H, Sotiriou C. Tumor infiltrating lymphocytes are prognostic in triple negative breast cancer and predictive for trastuzumab benefit in early breast cancer: results from the FinHER trial. Ann Oncol. 2014 Aug;25(8):1544-50. doi: 10.1093/annonc/mdu112. Epub 2014 Mar 7. PMID 24608200
- [Background] Salgado R, Denkert C, Demaria S, Sirtaine N, Klauschen F, Pruneri G, Wienert S, Van den Eynden G, Baehner FL, Penault-Llorca F, Perez EA, Thompson EA, Symmans WF, Richardson AL, Brock J, Criscitiello C, Bailey H, Ignatiadis M, Floris G, Sparano J, Kos Z, Nielsen T, Rimm DL, Allison KH, Reis-Filho JS, Loibl S, Sotiriou C, Viale G, Badve S, Adams S, Willard-Gallo K, Loi S; International TILs Working Group 2014. The evaluation of tumor-infiltrating lymphocytes (TILs) in breast cancer: recommendations by an International TILs Working Group 2014. Ann Oncol. 2015 Feb;26(2):259-71. doi: 10.1093/annonc/mdu450. Epub 2014 Sep 11. PMID 25214542
- [Background] Denkert C, von Minckwitz G, Brase JC, Sinn BV, Gade S, Kronenwett R, Pfitzner BM, Salat C, Loi S, Schmitt WD, Schem C, Fisch K, Darb-Esfahani S, Mehta K, Sotiriou C, Wienert S, Klare P, Andre F, Klauschen F, Blohmer JU, Krappmann K, Schmidt M, Tesch H, Kummel S, Sinn P, Jackisch C, Dietel M, Reimer T, Untch M, Loibl S. Tumor-infiltrating lymphocytes and response to neoadjuvant chemotherapy with or without carboplatin in human epidermal growth factor receptor 2-positive and triple-negative primary breast cancers. J Clin Oncol. 2015 Mar 20;33(9):983-91. doi: 10.1200/JCO.2014.58.1967. Epub 2014 Dec 22. PMID 25534375
- [Derived] Agarwal G, Vishvak Chanthar KMM, Katiyar S, Kumari N, Krishnani N, Sabaretnam M, Chand G, Mishra A, Lal P. Predictive and Prognostic Role of Tumor-Infiltrating Lymphocytes in Patients with Advanced Breast Cancer Treated with Primary Systemic Therapy. World J Surg. 2023 May;47(5):1238-1246. doi: 10.1007/s00268-023-06912-x. Epub 2023 Feb 3. PMID 36735048